CLINICAL TRIAL: NCT04714983
Title: A Phase I Safety and Window-of-opportunity Study of Preoperative Intratumoral Injection of OX40-ligand Expressing Oncolytic Adenovirus (DNX-2440) in Patients With Resectable Liver Metastasis
Brief Title: DNX-2440 for Resectable Colorectal Liver Metastasis
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: DNAtrix management decision not based on study design, safety, or site performance.
Sponsor: DNAtrix, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2440LM-002
Record Dates: First submitted 2020-12-09; First posted 2021-01-20 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Liver Metastases; Liver Metastasis Colon Cancer; Colorectal Cancer; Breast Cancer; Gastric Cancer; Periampullary Cancer; Melanoma; Renal Cell Cancer; Sarcoma; Squamous Cell Carcinoma; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Stomach Neoplasms; Melanoma; Carcinoma, Renal Cell; Sarcoma; Carcinoma, Squamous Cell; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose-level 1 (Experimental): The dose-level 1 arm will use a 3+3 design. A single dose of DNX-2440 will be delivered via intra-tumoral injection at Visit 1 and at Visit 3 (2 administrations in total) approximately 14 days apart.
  Interventions: Biological: DNX-2440
- Dose-level 2 (Experimental): The dose-level 2 arm will use a 3+3 design. A single dose of DNX-2440 will be delivered via intra-tumoral injection at Visit 1 and at Visit 3 (2 administrations in total) approximately 14 days apart.
  Interventions: Biological: DNX-2440
- Dose-level 3 (Experimental): The dose-level 3 arm will use a 3+3 design. A single dose of DNX-2440 will be delivered via intra-tumoral injection at Visit 1 and at Visit 3 (2 administrations in total) approximately 14 days apart.
  Interventions: Biological: DNX-2440

INTERVENTIONS:
Biological: DNX-2440 — DNX-2440 is a replication competent oncolytic adenovirus expressing human OX40 ligand.

SUMMARY:
The purpose of this study is to test an experimental oncolytic adenovirus called DNX-2440 in patients with resectable multifocal (≥ 2 lesions) liver metastasis, who are scheduled to have curative-intent liver resection surgery. Up to 18 patients will receive two sequential intra-tumoral injections of DNX-2440 into a metastatic liver tumor prior to surgery for liver resection, to evaluate safety and biological endpoints across 3 dose levels (dose escalation). Upon conclusion of the dose-escalation phase, the selected safe and biologically appropriate dose will be administered using the same schema for an additional 12 patients with colorectal cancer liver metastasis (expansion cohort) using established biologic endpoints.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged ≥ 18 years at time of consent
* Diagnosis of liver metastases from colorectal, breast, gastric, periampullary, melanoma, renal cell cancer, sarcoma, squamous cell carcinoma or gastrointestinal stromal tumor
* Multiple (≥ 2) liver tumors
* Candidate for curative-intent surgery
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Candidates eligible for targeted therapy, as per standard of care guidelines (and based on mutational status as indicated), must have completed therapy
* Preoperative chemotherapy is allowed

Key Exclusion Criteria:

* Recurrence of liver metastasis
* Diagnosis of neuroendocrine tumor liver metastasis
* Liver metastasis treated with > 12 cycles of systemic chemotherapy
* Condition that requires ongoing systemic immunosuppressive therapy
* Evidence of inadequate organ function based on lab parameters
* Liver transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) or total bilirubin > 5x the upper limits of normal
* Males or females who refuse to use a double-barrier form of birth control during the study and for up to 6 months after injection with DNX-2440

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) achieved during dose-escalation phase | 1.5 Years
  The MTD will be defined as the highest tolerated dose below the dose that results in greater than or equal to one-third of the subjects exposed who experience a dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Efficacy of DNX-2440 assessed by Tumor Regression Grade (TRG) score | 3 Years
  Efficacy in tumor cell killing will be measured using the TRG score (1-5) for the resected specimens
Viral replication | 3 Years
  Viral replication will be assessed by quantitative measurement of viral protein expression by IHC
Measure Immune response with cell response panels | 3 Years
  Immunotherapeutic responses will be assessed by examining features and measuring changes following the intervention for Immunologic microenvironment (T-cell and Myeloid-cell response panels-tissue).
Measure Immune response with ImmunoSEQsec | 3 Years
  Immunotherapeutic responses will be assessed by measuring changes in T-cell receptor (TCR) repertoire - tissue and blood.
Measure Immune response with ELISPOT | 3 Years
  Immunotherapeutic responses will be assessed by measuring T-cell response (ELISPOT - tissue/blood).

CONTACTS AND LOCATIONS:
Overall Officials: Joan Robbins, Ph.d, Study Director — DNAtrix, Inc.
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No